CLINICAL TRIAL: NCT04445259
Title: Study of the Treatment and Outcomes in Critically Ill Patients With COVID-19 and High Risk of Acute Kidney Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Sponsor
Other Study IDs: 283672
Record Dates: First submitted 2020-05-27; First posted 2020-06-24 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: COVID; Acute Kidney Injury; Critical Illness
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically Ill Patients with COVID-19: We plan to recruit patients who are admitted to intensive care units with COVID-19 diagnosis.

SUMMARY:
The aim is to describe the epidemiology and determine the independent risk factors for mortality and acute organ injury in AKI and to assess the impact of different treatment strategies on survival. This will allow the development of prevention strategies and design of appropriately powered intervention studies.

DETAILED DESCRIPTION:
Since the outbreak of coronavirus disease 2019 (COVID-19) began in December 2019 in China, over 1 million people have been infected and over 55,000 have died worldwide, and these numbers continue to rise. Combating this pandemic requires a multidisciplinary approach from the medical research community, including translational studies to understand the pathogenesis of disease, randomized controlled trials of novel and re-purposed pharmacotherapies, and rigorously conducted epidemiologic studies that include granular patient-level data.

Current knowledge of the clinical features and outcomes of COVID-19 is mostly limited to studies from China and Italy. In one of the larger such studies, which consisted of 1099 patients hospitalized in mainland China, only 173 (16%) were classified as having severe disease, and only 15 (1.4%) died. The study was therefore inadequately powered to determine independent risk factors for death. A larger study consisting of 72,314 patients was recently published by the Chinese Center for Disease Control and Prevention. This nationwide registry study identified several important findings, including the striking monotonic relationship between older age and greater risk of death. Important limitations of the study, however, were lack of granular patient-level data and relatively few patients (<5% of the cohort) who were critically ill. Among critically ill patients with COVID-19, acute mortality rates have been reported to be as high as 49-62%, underscoring the importance of studying this patient population. Data from the United Kingdom (UK) suggest that >50% of critically ill patients have a degree of acute kidney injury (AKI) and >20% need renal replacement therapy (RRT). Mortality is particularly high in those who are mechanically ventilated and need RRT (>75%).

Detailed information about the risk of AKI, contributing factors and reasons for high mortality in critically ill COVID-19 patients is lacking. To meet this urgent need, the investigators plan to collect clinical data from >250 critically ill patients with COVID-19 admitted to the intensive care unit (ICU) at Guy's & St Thomas' Hospital. The investigators will collaborate with Dr Gupta and Prof Leaf from Harvard Medical School, Boston (US) who are leading a similar study across >50 sites in the United States.

The aim is to describe the epidemiology and determine the independent risk factors for mortality and acute organ injury in AKI and to assess the impact of different treatment strategies on survival. This will allow the development of prevention strategies and design of appropriately powered intervention studies.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (aged ≥18 years)
2. Confirmed diagnosis of COVID-19
3. Hospitalized in the ICU for illness related to COVID-19
4. Any of the following:

   * Current in-patient in ICU
   * Previous in-patient in ICU and died in ICU or hospital
   * Previous in-patient in ICU and discharged from ICU alive

Exclusion Criteria:

1. Younger than 18 years old
2. On chronic dialysis within the last year or on dialysis at ICU admission
3. Functioning kidney transplant
4. No creatinine within 48 hours of ICU admission

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patients with confirmed diagnosis of COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-20 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of any stage of acute kidney injury | 14 days
  As defined by Kidney Diseases: Improving Global Outcomes (KDIGO) criteria

SECONDARY OUTCOMES:
Mortality | 14-day, hospital, and intensive care unit (ICU) mortality
  Mortality
Renal recovery | 14 days
  Defined by return of creatinine to < 1.5 times of baseline
Percentage of patients who receive renal replacement therapy | 14 days
  Percentage
Percentage of participants who are dialysis dependent | Through study completion, an average of 90 days
  Percentage of participants who are dialysis dependent
Free-days of vasoactive medications and mechanical ventilation | Day 30
  Days without vasoactive medications and mechanical ventilation
Length of intensive care unit and hospital stay | Through study completion, an average of 90 days
  Length of intensive care unit and hospital stay
Number of participants with consequences following AKI | Through study completion, an average of 90 days
  Congestive heart failure, Arrhythmia, Acute respiratory distress syndrome, Septic shock, Acute cardiac injury, pneumonia
Time from illness onset to need for mechanical ventilator support | Through study completion, an average of 30 days
  Time from illness onset to need for mechanical ventilator support

CONTACTS AND LOCATIONS:
Overall Officials: Nuttha Lumlertgul, MD, PhD, Principal Investigator — Guy's & St Thomas' Hospital
Locations (1):
- Guy's & St Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lumlertgul N, Baker E, Pearson E, Dalrymple KV, Pan J, Jheeta A, Weerapolchai K, Wang Y, Leach R, Barrett NA, Ostermann M. Changing epidemiology of acute kidney injury in critically ill patients with COVID-19: a prospective cohort. Ann Intensive Care. 2022 Dec 28;12(1):118. doi: 10.1186/s13613-022-01094-6. PMID 36575315
- [Derived] Lumlertgul N, Pirondini L, Cooney E, Kok W, Gregson J, Camporota L, Lane K, Leach R, Ostermann M. Acute kidney injury prevalence, progression and long-term outcomes in critically ill patients with COVID-19: a cohort study. Ann Intensive Care. 2021 Aug 6;11(1):123. doi: 10.1186/s13613-021-00914-5. PMID 34357478